CLINICAL TRIAL: NCT03574480
Title: Effectiveness of the Combined Use of Smartphone and Smartband Technology in the Improvement of Lifestyles in the Adult Population Over 65 Years of Age. Randomized Clinical Trial. EVIDENT Age Study
Brief Title: Smartphone Applications to Improve Lifestyles in Olders Over 65 Years
Acronym: EVIDENT-Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion y Formacion en Ciencias de la Salud (Other)
Collaborators: Instituto de Investigación Biomédica de Salamanca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: YB17/00003
Record Dates: First submitted 2018-06-20; First posted 2018-07-02 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2020-02

CONDITIONS: Telemedicine
Keywords: mHealth; Lifestyles; Elderly; Body composition; Cognitive performance; Quality of life
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): Advice on healthy diet and physical activity recommendations
  Interventions: Behavioral: Control (Advice on healthy diet and physical activity recommendations)
- Intervention (Experimental): * Advice on healthy diet and physical activity recommendations
  * Training for 3 months in use of a Smartphone application, designed to promote a healthy diet, increased physical acivity and decreased sedentary.
  Interventions: Behavioral: Intervention (training in use of a Smartphone application); Behavioral: Control (Advice on healthy diet and physical activity recommendations)

INTERVENTIONS:
Behavioral: Intervention (training in use of a Smartphone application) — The intervention group will be added a training for 3 months in use of a Smartphone application, designed to promote a healthy diet, increased physical acivity and decreased sedentary.
  Arms: Intervention
Behavioral: Control (Advice on healthy diet and physical activity recommendations) — Advice on healthy diet and physical activity recommendations

SUMMARY:
This is a randomized controlled clinical trial performed in urban primary care centers in Salamanca (Spain). Its objective is to evaluate the effect of an intervention based on the use of new information and communication technologies in a population of people over 65 years of age in the improvement of lifestyles, body composition, quality of life, cognitive performance and daily life activities.

DETAILED DESCRIPTION:
* Objective: To evaluate the effect of an intervention based on the use of new information and communication technologies in a population of people over 65 years of age.
* Design and setting: A randomized clinical trial of two parallel groups. Population: 140 participants over 65 years of age will be included, selected by consecutive sampling in primary care centers of Salamanca (Spain.
* Measurements and intervention: Lifestyles (physical activity, sedentarism and mediterranean diet), body composition, health-related quality of life, cognitive performance and daily life activities will be evaluated at 3 months. The advice on healthy diet and physical activity recommendations will be common to both groups. The intervention group will be added a training for 3 months in use of a Smartphone application, designed to promote a healthy diet, increased physical acivity and decreased sedentary.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed
* Age between 65 and 80 years

Exclusion Criteria:

* Cardiovascular disease
* Moderate or severe chronic obstructive pulmonary disease.
* Musculoskeletal disease that limits ambulation.
* Severe mental illness
* Score in the Mini-mental <24 points.
* Oncological disease in treatment.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Physical activity | 3 months
  Measurement by accelerometer (steps/day)

SECONDARY OUTCOMES:
Body composition | 3 months
  Measurement by Body fat percentage (%)
Cognitive performance | 3 months
  Measurement by MINI MENTAL STATE EXAMINATION (Score between 0 (Cognitive impairment) and 30 (normal))
Improve Quality of life | 3 months
  Measurement by the WHOQOL-AGE scale (Score between 13 (poor quality) and 65 (high quality))
Daily life activities | 3 months
  Measurement by PFEFFER FUNCTIONAL ACTIVITY Questionnaire (Score between 0 (normal) and 33 (Functional alteration))
Sedentarism | 3 months
  Measurement by Marshall questionnaire (sitting time - hours/day)
Adherence to the Mediterranean Diet | 3 months
  Measurement by the MEDAS scale (Score between 0 (poor adherence) and 14 (high adherence))

CONTACTS AND LOCATIONS:
Overall Officials: Jose I Recio-Rodriguez, PhD, Principal Investigator — University of Salamanca
Locations (1):
- Instituto Biosanitario de Salamanca. Research Unit La Alamedilla, Salamanca, Spain

REFERENCES:
- [Derived] Recio-Rodriguez JI, Gonzalez-Sanchez S, Tamayo-Morales O, Gomez-Marcos MA, Garcia-Ortiz L, Nino-Martin V, Lugones-Sanchez C, Rodriguez-Sanchez E. Changes in lifestyles, cognitive impairment, quality of life and activity day living after combined use of smartphone and smartband technology: a randomized clinical trial (EVIDENT-Age study). BMC Geriatr. 2022 Oct 6;22(1):782. doi: 10.1186/s12877-022-03487-5. PMID 36203135
- [Derived] Recio-Rodriguez JI, Lugones-Sanchez C, Agudo-Conde C, Gonzalez-Sanchez J, Tamayo-Morales O, Gonzalez-Sanchez S, Fernandez-Alonso C, Maderuelo-Fernandez JA, Mora-Simon S, Gomez-Marcos MA, Rodriguez-Sanchez E, Garcia-Ortiz L. Combined use of smartphone and smartband technology in the improvement of lifestyles in the adult population over 65 years: study protocol for a randomized clinical trial (EVIDENT-Age study). BMC Geriatr. 2019 Jan 23;19(1):19. doi: 10.1186/s12877-019-1037-y. PMID 30674284